CLINICAL TRIAL: NCT02805023
Title: Phase 1/2, Open Label & Double Blind Randomized Placebo-controlled Study to Assess the Feasibility of BGC101 (EnEPC) in the Treatment of Peripheral Arterial Disease (PAD) With Critical Limb Ischemia (CLI)
Brief Title: BGC101 (EnEPC) Autologous Cell Therapy From Patient's Own Blood for Treatment of Critical Limb Ischemia (CLI)
Acronym: EnEPC-CLI
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioGenCell Ltd. (Industry)
Collaborators: Laniado Hospital (Other); Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BioGenCell Ltd
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease; Peripheral Vascular Disease
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: the study will be double-blind for treatment allocation. Both BGC101 and placebo are supplied fresh in 5 mL ready-to use-syringes. Both BGC101 and placebo will be prepared by an unblinded trained personnel (external to the study staff members) who will not take part in the treatment and / or assessment of the patient. The patient will also be blinded and the investigator will delegate the unblinded and blinded staff in order to perform study procedures in a double-blind manner
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Intramuscular injection of control medium only
  Interventions: Biological: Control medium
- BGC101 (Experimental): Intramuscular injection of BGC101 (autologous EnEPC preparation)
  Interventions: Biological: BGC101 (autologous EnEPC preparation)

INTERVENTIONS:
Biological: BGC101 (autologous EnEPC preparation) — Intramuscular injections - single treatment session
  Arms: BGC101
Biological: Control medium — Intramuscular injections - single treatment session
  Arms: Placebo

SUMMARY:
Evaluate the feasibility of an autologous cell preparation composed of a mixture of cells enriched for endothelial progenitor cells (EnEPCs) and multipotent adult hematopoietic stem/progenitor cells (HSPC) (BGC101), in the treatment of patients suffering from peripheral arterial disease (PAD) with critical limb ischemia (CLI) who have not responded to optimal pharmacological treatment or control of risk factors and/or had a revascularization failure, and do not have the option of further revascularization treatment.

DETAILED DESCRIPTION:
BGC101 is designed to treat peripheral vascular disease in patients suffering from Critical Leg Ischemia (CLI) also referred to as chronic limb threatening ischemia (CLTI).

This part of the study is designed as a placebo double-blind randomized controlled trial (CRT) assessing the safety and efficacy of BGC101 in 45 eligible subjects in 2 Arms: Arm A: BGC101 treatment and Arm B: Placebo treatment. The Arm A:Arm B ratio is 2:1 A single dose treatment of the personalized cells by intramuscular injections into the affected leg takes less than 10 minutes.

Cells from a standard blood draw (with no pre-treatment, bone marrow aspiration, mobilization or apheresis) are transformed, within a day, into the investigational medicinal product BGC101.

BGC101, intended for autologous use, is a 'ready-to-use' cell suspension in prefilled syringes.

ELIGIBILITY:
Inclusion criteria:

1. Able to complete the study and comply with instructions.
2. Capable of understanding the purpose of the study and the contents of the informed consent form.
3. Aged at least 18 years.
4. Non-pregnant and non-lactating female patients.
5. Have the clinical indications diagnostic of CLI based on Rutherford category 4-5
6. Have at least one of the hemodynamic indicators of severe peripheral arterial occlusive disease (WIfI ischemia grade 2):

   * Toe pressure < 40 mmHg
   * Ankle pressure < 70 mmHg
   * TcPO2 < 40mmHg
7. Meeting one of the following conditions:

   1. Poor candidate for standard revascularization treatment for peripheral arterial disease due to unfavorable anatomy or high surgical/intervention risk based on the patient's underlying comorbidities.
   2. After undergoing clinically ineffective revascularization. Six weeks or more after undergoing a prior index limb revascularization the patient demonstrates:

      * No improvement in clinical signs and symptoms of CLI as evidenced by lack of improvement in rest pain (when not under increased pain relief) and/or inadequate wound healing or progression of tissue loss despite adequate standard treatment.
      * Ongoing ischemia as defined above in the inclusion criterion 6.
      * The patient is no longer amenable to further interventional or surgical revascularization (see inclusion criterion 7c below).
   3. Four weeks or more after a revascularization failure.

      * Technical Failure of the revascularization (inability to successfully cross or treat the intended target arterial path, thrombosis of the bypass graft or treated artery within 7 days of procedure)
      * Hemodynamic Failure of the revascularization (lack of improvement in toe pressure, ankle pressure, or TcPO2) post-procedure

Exclusion criteria:

1. Severe uncorrected aorto-iliac and/or common femoral artery disease, absent of femoral pulse or monophasic common femoral artery Doppler waveform.
2. Concurrent therapy that, in the Investigator's opinion, would interfere with the evaluation of the feasibility of the study medication.
3. Treatment with any investigational product within the last 6 months or enrollment in any active study involving the use of investigational devices or drugs.
4. Presence of any other condition or circumstance that, in the judgment of the investigator, might negatively impact the outcomes of the treatment under investigation.
5. Prognosis of a major amputation (below or above the knee), within 4 weeks after screening.
6. Severe wound (WIfI wound grade 2 or 3).
7. Significant ongoing infection (WIfI infection grade 2 or 3).
8. Relative or absolute contraindications for intramuscular injections at the intended treatment site, in cases such as severe skin lesions, severe edema or morbid obesity, based on clinician opinion.
9. Patient suffering from active vasculitis
10. Blood transfusions during the preceding 4 weeks (to exclude the potential of non-autologous cells in the harvested blood).
11. Hemoglobin (Hb) less than 9 g/dL.
12. Patient with HbA1C > 8.5%
13. Myocardial infarction, cerebral infarction , uncontrolled myocardial ischemia or persistent severe heart failure (ejection fraction [EF] < 25%) during the preceding 3 months.
14. Heart failure (New York Heart Association [NYHA] 3-4).
15. Significant valvular disease or less than 4 weeks after valve replacement or repair
16. Renal failure (estimated glomerular filtration rate [eGFR] < 30 mL/min/1.73 m², chronic kidney damage stage 4-5).
17. Liver failure, Model for End-stage Liver Disease (MELD) scores 15 and higher.
18. Liver function tests more than three times normal upper limit (normal limits being defined in each local laboratory) (glutamic-oxaloacetic transaminase [GOT], glutamic-pyruvic transaminase [GPT], alkaline phosphatase [AlkP], gamma-glutamyl transferase [GGT], lactate dehydrogenase [LDH]).
19. Abnormal coagulation tests when not under warfarin (normalized prothrombin time [PT INR] >2).
20. Pregnant or lactating women at entry of study.
21. People who are unwilling to agree to use acceptable methods of contraception during the study.
22. Malignancy within the preceding 3 years, except basal cell carcinoma.
23. Concurrent acute infectious disease with septicemia
24. Chronic infectious disease (human immunodeficiency virus-1 [HIV-1], human immunodeficiency virus-2 [HIV-2], hepatitis B virus [HBV], hepatitis C virus [HCV]).
25. Immunodeficiency syndrome.
26. Raynaud's syndrome
27. Systemic treatment with cytotoxic and/or immunosuppressive treatment.
28. Inability to communicate (that may interfere with the clinical evaluation of the patient).
29. Patient unlikely to be available for follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety (Incidence of adverse events) | 12 Months
  * Incidence and proportion of incidence between treatment arms of adverse events of specific interest (AESI) and injection-related AE
  * Incidence of serious adverse events (SAEs) including SAEs related or probably related to the treatment
  * Vital signs, physical examination, and electrocardiogram (ECG)
  * Safety laboratory values of hematology, blood chemistry, and urinalysis
  * Local tolerability (injection site reaction)
Efficacy (Improvement of indication signs) | 12 Months
  * Major amputation (below or above the knee) rate at Month 12
  * Major amputation-free survival (AFS) rate at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo J Baytner, MD, Principal Investigator — Director of Vascular Surgery, Laniado Hospital, IL; Michael Conte, MD, Principal Investigator — University of California, San Francisco - Division Vascular and Endovascular surgery; Edouard Aboian, MD, Principal Investigator — Yale University School of Medicine- Division of Vascular Surgery, Department of Surgery; Caitlin Hicks, MD, Principal Investigator — Division of Vascular Surgery and Endovascular Therapy, Johns Hopkins Hospital; Tony Karram, MD, Principal Investigator — Director Department of Vascular Surgery & Transplantation Rambam Health Care Campus - IL; Nathalie Moreels, MD, Principal Investigator — University Hospital Ghent-Thoracale en vasculaire heelkunde; Jeffrey J Siracuse, MD, Principal Investigator — Boston Medical Center; Khanjan Nagarsheth, MD, Principal Investigator — University of Maryland; Paata Meshveliani, MD, Principal Investigator — West Georgia Medical Center (Kutaisi Hospital); Moshe Halak, MD, Principal Investigator — The Sheba Fund for Health Services and Research, Sheba Medical Center at Tel HaShomer; Igor Laskowski, MD, Principal Investigator — New York Medical College ("NYMC") and Westchester County Health Care Corporation, operator of Westchester Medical Center.; Mark Wyers, MD, Principal Investigator — Beth Israel Deaconess Medical Center (Harvard-Boston); Alisha Oropallo, MD, Principal Investigator — Northwell Health; Alexander Reyzelman, MD, Principal Investigator — Center for Clinical Research Castro Valley- Main site Post Street -Satellite site
Locations (5):
- United States (3):
  - University of San Francisco, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Johns Hopkins Hospital, Baltimore, Maryland
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Laniado Hospital, Netanya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Porat Y, Assa-Kunik E, Belkin M, Krakovsky M, Lamensdorf I, Duvdevani R, Sivak G, Niven MJ, Bulvik S. A novel potential therapy for vascular diseases: blood-derived stem/progenitor cells specifically activated by dendritic cells. Diabetes Metab Res Rev. 2014 Oct;30(7):623-34. doi: 10.1002/dmrr.2543. PMID 24638886